CLINICAL TRIAL: NCT05234242
Title: Inguinal Hernia Treatment: Stationary/Inpatient vs. Ambulatory/Outpatient Setting - HerStAmb Study (Prospective Non-randomized Multicenter Comparative Study)
Brief Title: Inguinal Hernia Treatment: Stationary/Inpatient vs. Ambulatory/Outpatient Setting - HerStAmb Study
Status: Completed | Type: Observational
Sponsor: Dr. Michal Ziga (Other)
Responsible Party: Sponsor-Investigator, Dr. Michal Ziga, Dr., Cantonal Hospital Schaffhausen
Organization: Cantonal Hospital Schaffhausen (Other)
Other Study IDs: HerStAmb Study
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Outcome of Outpatient/Ambulatory and Inpatient/Stationary Setting
Keywords: inguinal hernia treatment, AVOS, complications, re-admission, outcome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- stationary/inpatient
  Interventions: Procedure: inguinal hernia repair
- ambulatory/outpatient
  Interventions: Procedure: inguinal hernia repair

INTERVENTIONS:
Procedure: inguinal hernia repair — inguinal hernia repair performed either in stationary/inpatient or ambulatory/outpatient setting

SUMMARY:
Since 01/2018, AVOS (ambulant vor stationär = ambulatory to stationary) regulation has been progressively implemented in hospitals across Switzerland for certain surgical procedures, including the treatment of inguinal hernias.

The aim of this prospective, non-randomized, multicenter study was to compare the outcome of outpatient/ambulatory and inpatient/stationary postoperative care by examining the re-admission rate, complication rate and quality of life in patients with primary unilateral inguinal hernia repair.

DETAILED DESCRIPTION:
Inguinal hernia repair procedures are among the most performed surgeries worldwide, with more than 20 million people undergoing the procedure annually. Various tension or tension-free operation-techniques have been developed over the years. According to the International Guidelines developed by HerniaSurge Group in 2018, the gold standard are tension-free procedures with prosthetic material (mesh), either laparoscopic (total extraperitoneal patch (TEP), transabdominal preperitoneal patch (TAPP) or open surgery (Lichtenstein). In Switzerland, open surgery is used for 58.5% of hernias while 41.5% are operated on laparoscopically with the TEP as the first choice. Similar data is also reported in Great Britain. The development of modern anaesthesia as well as the safe techniques performed by experienced surgeons permit treatment of inguinal hernias in the outpatient setting, while the American Society of Anaesthesiologists (ASA) state that I - III class patients who have satisfactory care at home should be considered for day surgery. A crucial role in the process is played by the anaesthesiologist and surgeon who are responsible for perioperative management and the early postoperative phase. The factors in favour or against the suitability of day surgery include environmental factors (hospital, physician) as well as patient-related factors and thus a tailored approach must be considered for each patient. Outpatient treatment can only be performed in a hospital with suitable infrastructure (pre-assessment, day surgery department) and a high caseload, which usually results in the surgery being routine, with less complications occurring and a shorter procedure time. Control of postoperative pain and nausea are also very important for quick discharge. The financial support of the healthcare system also plays a significant role.

While there is a growing trend towards day surgery, considerable variations exist internationally and between hospitals at the national level. The evaluation of the French hernia register by Drissi et al showed slightly lower re-admission rate in ambulatory patients while Steger et al report a positive experience as well as acceptance of the ambulatory TEP procedure in one centre in Germany. Köckerling et al showed no significant differences in pain and recurrence rate in primary elective unilateral inguinal hernia treated in the outpatient setting. However, there are no prospective studies and data comparing outpatient/ambulatory vs. inpatient/stationary treatment setting in respect of complications, re-admission rate and patient outcome/quality of life.

Since 01/2018, AVOS (ambulant vor stationär = ambulatory to stationary) regulation has been progressively implemented in Swiss hospitals for certain procedures - inguinal hernia treatment included. AVOS regulation passed into law in 01/2019, with small modifications made to the recommendations of the European Hernia Society for hernia treatment in the outpatient setting.

Our study is the first prospective study comparing the efficiency and the effectiveness of ambulatory/outpatient and stationary/inpatient postoperative management through the investigation of the postoperative re-admission rate, complication rate and patient outcome/quality of life after the procedure in a group of patients with primary unilateral inguinal hernia.

The study was designed as a prospective non-randomized multicentre study carried out at 2 Swiss hospitals (Centre A: Triemli City Hospital, Centre B: Cantonal Hospital Schaffhausen) between 01/2019 - 04/2020 following the same study protocol. All patients were seen preoperatively in an outpatient clinic or emergency room. Patients were examined by a surgeon and anesthesiologist and after evaluation of the objective status, comorbidities and social situation, the procedure and postoperative management according to the AVOS guidelines were decided. Patients with a recurrent or bilateral hernia were excluded as they could bias the re-admission rate as the complication rate and need for analgesia are higher in these patients. The primary endpoint of the study was re-admission rate within 6 weeks postoperatively due to complication (a: seroma, b: hematoma, c: wound infection/dehiscence, d: recurrence, e: pain, f: postop. delirium). Secondary endpoints were the complication rate and patient outcome at 6 weeks postoperatively measured by the SF-36 questionnaire, a well-established tool for measuring the performance status and quality of life of patients in 8 different categories.

Intention-to-treat analysis was done and descriptive statistics using the chi-square test for categorical variables was used to measure the relationship between treatment setting and complication rate as well as treatment setting and re-admission rate. Per protocol analysis with an independent t-test was used to find any significant difference between the treatment setting and mean clinical outcome of the patients measured by SF-36 at 6 weeks postoperatively. P < 0.05 was statistically significant. The study was approved by the Ethics Committee of Zürich (Kantonale Ethikkomission Zürich, BASEC Nr. 2018-10832)

ELIGIBILITY:
Inclusion Criteria:

1. Primary unilateral inguinal hernia
2. Written informed consent after participants' information,
3. Outpatient or inpatient treatment

Exclusion Criteria:

1. Recurrent hernia
2. Bilateral hernia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients included in the study were diagnosed with the symptomatic primary unilateral inguinal hernia. They have various jobs and different lifestyles.
Sampling Method: Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
re-admission rate | 6 weeks
complication rate | 6 weeks
  a: seroma, b: hematoma, c: wound infection/dehiscence, d: recurrence, e: pain, f: postop. delirium
quality of life | 6 weeks
  SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michal Ziga, Dr., Principal Investigator — Cantonal Hospital Schaffhausen
Locations (1):
- Cantonal Hospital Schaffhausen, Schaffhausen, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ziga M, Burla L, Imhof A, Gurtler T, Weber M. Inguinal hernia treatment in Switzerland: inpatient vs. outpatient setting - HerStAmb Study (prospective observational two-centre comparative study). Langenbecks Arch Surg. 2023 Jan 9;408(1):14. doi: 10.1007/s00423-023-02766-y. PMID 36622458